CLINICAL TRIAL: NCT03225300
Title: Evaluation the Prognostic Significance of High Radiation Dose in Malignant Glioma Patients Treated With Chemoradiation
Brief Title: Simultaneous Integrated Boost in Malignant Glioma Patients Treated With Chemoradiation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE17194B
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Glioblastoma Multiforme; Chemoradiation
Keywords: Glioblastoma; Chemoradiation; Simultaneous integrated boost
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: A prospectively single arm in single institution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simultaneous integrated boost (Experimental): In this protocol, the newly diagnosed, primary glioblastoma patients receive SIB 69 Gy/30 fractions to preoperative tumor bed and surgical cavity, while 60 Gy/30 fractions were covering preoperatively edematous area. PTV is 5 mm.
  Interventions: Radiation: Simultaneous integrated boost

INTERVENTIONS:
Radiation: Simultaneous integrated boost — Simultaneous integrated boost (SIB), a field-in-field escalation technique, has been introduced to deliver higher radiation dose to the certain part of target with the same fractionation scheme.

SUMMARY:
Simultaneous integrated boost (SIB), a field-in-field escalation technique, has been introduced to deliver higher radiation dose to the certain part of target with the same fractionation scheme. The aim of this study was to investigate the value of chemoradiation (CCRT) using SIB in glioblastoma and the correlation with surgical extent.

DETAILED DESCRIPTION:
The SIB technique provides the higher radiobiological effect with the same fractionation scheme, i.e. 69 Gy over 6 weeks, which might increase the loco-regional control. Besides, the co-registration with magnetic resonance imaging (MRI) strengthens the precision of target delineation as well as higher possibility to spare adjacent normal brain tissue.

In this protocol, the newly diagnosed, primary glioblastoma patients received SIB 69 Gy/30 fractions to preoperative tumor bed and surgical cavity, while 60 Gy/30 fractions were covering preoperatively edematous area. To determine the status of surgical extent, postoperative CT scan and MRI was acquired within 72 hours and at 4th week after surgery. During the period of chemoradiation, acute neurotoxicity and hematological toxicity was assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* newly diagnosed, tissue-proven glioblastoma
* pre-radiotherapy Karnofsky performance score (KPS) ≧60.

Exclusion Criteria:

* any previous history of chemotherapy or radiotherapy
* receiver of any investigating agents
* recurrent GBM
* any second malignancies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free survival rate | at the end of first year
  Actual one-year progression-free survival rate

SECONDARY OUTCOMES:
Surgical extent | CT within 72 hours and MRI at 4th week after surgery
  No contrast-enhanced area: gross total resection; Any contrast-enhanced area: residual tumor

CONTACTS AND LOCATIONS:
Overall Officials: Weir Chiang You, M.D. Ph.D., Study Chair — Dempartment of Radiation Oncology
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Bauchet L, Mathieu-Daude H, Fabbro-Peray P, Rigau V, Fabbro M, Chinot O, Pallusseau L, Carnin C, Laine K, Schlama A, Thiebaut A, Patru MC, Bauchet F, Lionnet M, Wager M, Faillot T, Taillandier L, Figarella-Branger D, Capelle L, Loiseau H, Frappaz D, Campello C, Kerr C, Duffau H, Reme-Saumon M, Tretarre B, Daures JP, Henin D, Labrousse F, Menei P, Honnorat J; Societe Francaise de Neurochirurgie (SFNC); Club de Neuro-Oncologie of the Societe Francaise de Neurochirurgie (CNO-SFNC); Societe Francaise de Neuropathologie (SFNP); Association des Neuro-Oncologues d'Expression Francaise (ANOCEF). Oncological patterns of care and outcome for 952 patients with newly diagnosed glioblastoma in 2004. Neuro Oncol. 2010 Jul;12(7):725-35. doi: 10.1093/neuonc/noq030. Epub 2010 Apr 2. PMID 20364023
- [Background] Monjazeb AM, Ayala D, Jensen C, Case LD, Bourland JD, Ellis TL, McMullen KP, Chan MD, Tatter SB, Lesser GJ, Shaw EG. A phase I dose escalation study of hypofractionated IMRT field-in-field boost for newly diagnosed glioblastoma multiforme. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):743-8. doi: 10.1016/j.ijrobp.2010.10.018. Epub 2011 Jan 13. PMID 21236604